CLINICAL TRIAL: NCT04019184
Title: Biomarker-guided Implementation of Glutamine to Reduce the Occurence of AKI After Cardiac Surgery
Brief Title: Reduction of Occurence of Acute Kidney Injury (AKI) Through Administration of Glutamine
Acronym: Glacé
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital Muenster (Other)
Collaborators: Fresenius Kabi (Industry); IZKF (Interdisciplinary Centre for Clinical Research (IZKF), Muenster) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UKM17_0035; 2018-002832-25 (EudraCT Number)
Record Dates: First submitted 2019-07-04; First posted 2019-07-15 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Cardiac Surgery; Acute Kidney Injury
Keywords: Cardiac surgery; glutamine
MeSH Terms: conditions — Acute Kidney Injury | interventions — alanylglutamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glutamine group (Experimental): Intravenous infusion of 0.5 g/kg body weight (2.5 ml/kg body weight) L-alanyl-Lglutamine over 12 h after randomization
  Interventions: Drug: L-Alanyl/L-Glutamine
- Control group (Placebo Comparator): Intravenous infusion of 2.5 ml/kg body weight sodium chloride 0.9 % over 12 h after randomization
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: L-Alanyl/L-Glutamine — Immediately after randomization (not longer than 30 min after fulfilling eligibility criteria), patients will receive intravenous infusions with the investigational drug
  Arms: Glutamine group
Drug: Placebo — Immediately after randomization (not longer than 30 min after fulfilling eligibility criteria), patients will receive intravenous infusions with the placebo
  Arms: Control group

SUMMARY:
The aim of this study is to evaluate whether the application of glutamine versus control in patients with high risk for AKI identified by biomarkers can reduce kidney damage after cardiac surgery.

DETAILED DESCRIPTION:
Cardiac surgery is characterized by an increased production of free radicals as a consequence of surgical trauma, ischemia-reperfusion injury, inflammatory response syndrome in response to the use of the extracorporeal circulation. This results in an increased production and release of free radicals which may lead to an exhaustion of antioxidants and organ failure since the lungs, kidneys, liver and gastrointestinal tract are particularly susceptible to reactive oxidant species. Glutamine is considered as a conditionally indispensable amino acid in catabolic states of critically ill patients. It belongs, together with other mediators, to the host defense as major intracellular direct free radical scavengers. Its depletion has been demonstrated to be an independent predictor of mortality in a group of ICU (intensive care unit) patients. Clinical studies showed a positive outcome effect. In animal models, glutamine reduces the occurrence of AKI after ischemia-reperfusion injury. This could be demonstrated through reduced functional markers as well as reduced renal biomarker levels. Preliminary data suggest that glutamine has pleiotropic effects since it has effects on the immune system (reduced expression of cytokines) as well as on tubular epithelial cells (unpublished animal data from our laboratory).

Thus, a randomized-controlled trial to analyze the effects of glutamine supplementation in high risk patients identified by renal biomarkers undergoing cardiac surgery with cardiopulmonary bypass (CPB) on the effects of kidney damage is urgently needed.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing cardiac surgery with CPB
* Urinary [TIMP-2]*[IGFBP7] >= 0.3 4h after CPB
* Written informed consent

Exclusion Criteria:

* Preexisting AKI (stage 1 and higher)
* Patients with cardiac assist devices
* Pregnant women, nursing women and women of childbearing potential
* Known (Glomerulo-) Nephritis, interstitial nephritis or vasculitis
* Chronic kidney disease (CKD) with estimated glomerular filtration rate (eGFR) < 30 ml/min
* Dialysis dependent CKD
* Prior kidney transplant within the last to 12 months
* Hypersensitivity to the active substance, or to any of the excipients of the study medication
* Hepatic insufficiency
* Severe metabolic acidosis (pH < 7.2)
* Participation in another intervention trial in the past 3 months
* Persons with any kind of dependency on the investigator or employed by the institution responsible or investigator
* Persons held in an institution by legal or official order

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2019-07-18 (Actual); Primary Completion 2020-02-13 (Actual); Study Completion 2020-05-13 (Actual)

PRIMARY OUTCOMES:
Kidney damage after cardiac surgery identified by measuring biomarkers ([TIMP-2]*[IGFBP7] | 12 hours after cardiac surgery
  The presence of tissue inhibitor of metalloproteinases (TIMP-2) and insulin-like grwoth-factor binding protein 7 (IGFBP7) in the urine will be measured.

SECONDARY OUTCOMES:
Occurence of acute kidney injury according to the KDIGO (Kidney Disease: Improving Global Outcomes) criteria | 72 hours after end of cardiac surgery
Severity of acute kidney injury (number of patients with KDIGO stage 1, KDIGO stage 2 or KDIGO stage 3) | 72 hours after end of cardiac surgery
  Definition and classification of acute injury according to the KDIGO (Kidney Disease Improving Global Outcomes) clinical practice guidelines on acute kidney injury
Creatinine Clearance | one day after cardiac surgery
Free-days of vasoactive medications and mechanical ventilation | 28 days after cardiac surgery
Renal recovery | 30 days after cardiac surgery
  Renal recovery is defined as serum creatinine levels < 0.5 mg/dL higher than baseline serum creatinine
Renal recovery | 60 days after cardiac surgery
  Renal recovery is defined as serum creatinine levels < 0.5 mg/dL higher than baseline serum creatinine
Renal recovery | 90 days after cardiac surgery
  Renal recovery is defined as serum creatinine levels < 0.5 mg/dL higher than baseline serum creatinine
Mortality | 30 days after cardiac surgery
Mortality | 60 days after cardiac surgery
Mortality | 90 days after cardiac surgery
ICU and Hospital stay | up to 90 days after cardiac surgery (until discharge)
Number of patients with renal replacement therapy | up to 90 days after cardiac surgery

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Zarbock, MD, PhD, Principal Investigator — University Hospital Muenster, Dept. of Anesthesiology, Intensive Care and Pain Medicine
Locations (1):
- University Hospital Münster, Münster, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Weiss R, Meersch M, Gerke M, Wempe C, Schafers M, Kellum JA, Zarbock A. Effect of Glutamine Administration After Cardiac Surgery on Kidney Damage in Patients at High Risk for Acute Kidney Injury: A Randomized Controlled Trial. Anesth Analg. 2023 Nov 1;137(5):1029-1038. doi: 10.1213/ANE.0000000000006288. Epub 2022 Nov 29. PMID 36730070